CLINICAL TRIAL: NCT00831753
Title: Immunogenicity Study of DTaP-IPV-Hep B-PRP~T Combined Vaccine in Comparison to Infanrix®Hexa, at 2-4-6 Months of Age in Healthy Peruvian Infants
Brief Title: Study of DTaP-IPV-Hep B-PRP~T Combined Vaccine Compared to Infanrix®Hexa in Healthy Peruvian Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A3L17
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Haemophilus Influenzae Type b; Hepatitis B
Keywords: Diphtheria; Tetanus; Pertussis; whooping cough; Haemophilus influenzae type b; Hepatitis B; Poliomyelitis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Haemophilus Infections; Hepatitis B; Poliomyelitis | interventions — DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): DTaP-IPV-Hep B-PRP~T vaccine group
  Interventions: Biological: DTaP IPV HB PRP~T vaccine
- Group 2 (Active Comparator): Infanrix® Hexa vaccine group
  Interventions: Biological: DTaP-HB-IPV and Haemophilus influenzae type b

INTERVENTIONS:
Biological: DTaP IPV HB PRP~T vaccine — 0.5 mL, Intramuscular
  Arms: Group 1
Biological: DTaP-HB-IPV and Haemophilus influenzae type b — 0.5 mL, Intramuscular
  Other Names: Infanrix® Hexa
  Arms: Group 2

SUMMARY:
The study aims to confirm that, in Peruvian infants, the investigational DTaP-IPV Hep B-PRP~T vaccine has immunological and safety profiles that are comparable to those of the control vaccine that is already marketed (Infanrix®Hexa)

Primary Objective:

To demonstrate that the hexavalent DTaP-IPV-Hep B-PRP~T combined vaccine induces an immune response that is at least as good as the response following Infanrix®Hexa in terms of seroprotection rates to HB, one month after a three-dose primary series (2, 4 and 6 months)

Secondary Objectives:

* To describe in each group the immunogenicity to vaccine components (for DTaP-IPV-Hep B-PRP~T and Infanrix®Hexa) one month after the third dose of the primary series.
* To assess the overall safety in each group one month after each dose of the primary series and through the entire study.

DETAILED DESCRIPTION:
The present trial will involve two-month old Peruvian infants, randomly assigned to receive three doses of either the investigational or the control vaccine at 2, 4, and 6 months of age.

ELIGIBILITY:
Inclusion Criteria :

* Two month old infant (50 to 71 days old) on the day of inclusion, of either gender
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg
* Mother negative for Hepatitis B surface Antigen (HBsAg) in approximately the last 30 days of pregnancy (≥ 36 weeks of amenorrhea) or in the 30 days post partum
* Informed consent form signed by both parents. If one or both parent(s) are under 18 years of age, the subject's grandparent(s) should also sign. An independent witness should also sign if the parent(s)/grandparent(s) are illiterate
* Able to attend all scheduled visits and to comply with all trial procedures
* Received Bacillus Calmette Guerin (BCG) vaccine between birth and one month of life in agreement with the national immunization calendar.

Exclusion Criteria :

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to the trial vaccine or a vaccine containing the same substances
* Congenital or acquired immunodeficiency, or immunosuppressive therapy such as long-term (for more than 2 weeks) systemic corticosteroid therapy within the last four weeks
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received since birth
* Any vaccination in the 4 weeks preceding the first trial vaccination
* Any planned vaccination during the trial (until Visit 06), except the study vaccines, rotavirus vaccine and pneumococcal conjugate vaccines
* Documented history of pertussis, tetanus, diphtheria, poliomyelitis, hepatitis B or Haemophilus influenzae type b infection(s) (confirmed either clinically, serologically, or microbiologically)
* Previous vaccination against pertussis, tetanus, diphtheria, poliomyelitis, hepatitis B or Haemophilus influenzae type b infection(s)
* Known personal or maternal history of Human Immunodeficiency Virus, hepatitis B or hepatitis C seropositivity
* Known thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination
* History of seizures
* Febrile (temperature ≥ 38.0°C) or acute illness on the day of inclusion.

Ages: 50 Days to 71 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 263 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Lima, Peru

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 23 May 2008 to 18 July 2008 at 1 clinical center in Peru.
Pre-assignment Details: A total of 263 participants who met the inclusion and exclusion criteria were randomized and vaccinated in the study.
Groups:
- DTaP-IPV-Hep B-PRP~T Group: All participants received a 3-dose primary series of diphtheria, tetanus, pertussis (2-component acellular), recombinant hepatitis B (Hep B) Hansenula polymorpha and inactivated poliomyelitis vaccine (IPV) adsorbed, and Haemophilus influenzae type b (Hib) vaccine, polyribosyl ribitol phosphate conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T) combined vaccine. A dose at 2, 4, and 6 months of age, respectively.
- Infanrix Hexa™ Group: All participants received a 3-dose primary series of Infanrix hexa™ vaccine, with 1 dose each at 2, 4, and 6 months of age, respectively.
Period: Overall Study
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | Infanrix Hexa™ Group
Started | 132 | 131
Completed | 132 | 131
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | Infanrix Hexa™ Group | Total
Number analyzed (Participants) | 132 | 131 | 263
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 132 | 131 | 263
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 1.75 (0.132) | 1.72 (0.123) | 1.74 (0.128)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 74 | 132
  Male | 74 | 57 | 131
Region of Enrollment [Number; unit: Participants]
  Peru | 132 | 131 | 263

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Seroprotection for Anti Hep-B After a Primary Series of Vaccination With Either DTaP-IPV-Hep B-PRP~T or Infanrix Hexa™
Description: Anti-hepatitis B (Hep B) antibodies were measured by chemiluminescence detection. Seroprotection was defined as a titer ≥ 10 mIU/mL.
Time Frame: Day 150 (1 month after dose 3)
Population: Seroprotection against Hep B was assessed in all participants who did not have any protocol violation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | Infanrix Hexa™ Group
Number analyzed (Participants) | 132 | 130
Participants | 131 | 130 [0 to 0]

2. Primary Outcome: Number of Participants Achieving Seroprotection to Vaccine Antigens After a Primary Series Vaccination With Either DTaP-IPV-Hep B-PRP~T or Infanrix Hexa™ Vaccine.
Description: Antibody titers were measured by chemiluminescence detection for hepatitis B (Hep B), by Farr type radioimmunoassay for Haemophilus influenzae type b (PRP), and by toxin neutralization test for diphtheria. Seroprotection criteria were defined as:
  Criteria 1: Anti-Hep B titer ≥ 10 mIU/mL; Anti-PRP titer ≥ 0.15 µg/mL; Anti-diphtheria titer ≥ 0.01 IU/mL.
  Criteria 2: Anti-Hep B titer ≥ 100 mIU/mL; Anti-PRP titer ≥ 1 µg/mL; Anti-diphtheria titer or ≥ 0.1 IU/mL.
Time Frame: Day 150 (1 month after dose 3)
Population: Seroprotection was assessed in all participants who did not have any protocol violation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | Infanrix Hexa™ Group
Number analyzed (Participants) | 132 | 130
Participants
  Anti-Hep B (Criteria 1) | 131 | 130 [0 to 0]
  Anti-Hep B (Criteria 2) | 124 | 129 [0 to 0]
  Anti-PRP (Criteria 1) | 132 | 129 [0 to 0]
  Anti-PRP (Criteria 2) | 112 | 109 [0 to 0]
  Anti-Diphtheria (Criteria 1) | 126 | 130 [0 to 0]
  Anti-Diphtheria (Criteria 2) | 77 | 85 [0 to 0]

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies to Vaccine Antigens After a Primary Series of Vaccination With Either DTaP-IPV-Hep B-PRP~T or Infanrix Hexa™ Vaccine.
Description: Antibody titers were measured by chemiluminescence detection for hepatitis B (Hep B), by Farr type radioimmunoassay for Haemophilus influenzae type b (PRP), and by toxin neutralization test for diphtheria.
Time Frame: Day 150 (1 month after dose 3)
Population: Antibody GMTs were assessed in all participants who did not have any protocol violation that might have interfered with primary criteria evaluation (Per-Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | Infanrix Hexa™ Group
Number analyzed (Participants) | 132 | 130
Titers (1/dilutions)
  Anti Hep B | 986 [764 to 1270] | 1139 [961 to 1350]
  Anti PRP | 5.22 [4.04 to 6.73] | 3.93 [3.17 to 4.89]
  Anti Diphtheria | 0.156 [0.119 to 0.204] | 0.192 [0.154 to 0.239]

4. Secondary Outcome: Number of Participants Reporting Solicited Injection Site or Solicited Systemic Reactions After Vaccination With Either DTaP-IPV-Hep B-PRP~T or Infanrix Hexa™ Vaccine.
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling. Solicited Systemic Reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia, Irritability.
  Grade 3 reactions were defined as: Pain, cries when injected limb is moved or movement of injected limb is reduced; Erythema and Swelling ≥ 5 cm; Pyrexia > 39.5ºC; Vomiting ≥ 6 episodes per 24 hour or requiring parenteral hydration; Crying, > 3 hours; Somnolence, sleeping most of the time or difficult to wake up; Anorexia refuses ≥ 3 feeds/meals or refuses most feeds/meals; Irritability inconsolable.
Time Frame: Day 0 up to Day 7 after each injection
Population: Solicited reactions were assessed in all participants who received at least one dose of investigational or control vaccine, according to the vaccine actually received (Safety Analysis Population).
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | Infanrix Hexa™ Group
Number analyzed (Participants) | 132 | 131
Participants
  Pain Post Injection 1 | 82 | 71 [0 to 0]
  Pain Post Injection 2 | 68 | 68 [0 to 0]
  Pain Post Injection 3 | 53 | 55 [0 to 0]
  Grade 3 Pain Post Any Injection | 10 | 6 [0 to 0]
  Erythema Post Injection 1 | 32 | 16 [0 to 0]
  Erythema Post Injection 2 | 48 | 30 [0 to 0]
  ErythemaPost Injection 3 | 45 | 46 [0 to 0]
  Grade 3 Erythema Post Any Injection | 3 | 5 [0 to 0]
  Swelling Post Injection 1 | 34 | 12 [0 to 0]
  Swelling Post Injection 2 | 26 | 24 [0 to 0]
  Swelling Post Injection 3 | 28 | 32 [0 to 0]
  Grade 3 Swelling Post Any Injection | 3 | 2 [0 to 0]
  Pyrexia Post Injection 1 | 11 | 11 [0 to 0]
  Pyrexia Post Injection 2 | 21 | 17 [0 to 0]
  Pyrexia Post Injection 3 | 18 | 18 [0 to 0]
  Gade 3 Pyrexia Post Any Injection | 0 | 3 [0 to 0]
  Any Vomiting Post Injection 1 | 20 | 24 [0 to 0]
  Any Vomiting Post Injection 2 | 8 | 6 [0 to 0]
  Vomiting Post Injection 3 | 6 | 10 [0 to 0]
  Grade 3 Vomiting Post Any Injection | 0 | 0 [0 to 0]
  Crying Post Injection 1 | 81 | 68 [0 to 0]
  Crying Post Injection 2 | 57 | 52 [0 to 0]
  Crying Post Injection 3 | 43 | 47 [0 to 0]
  Grade 3 Crying Post Any Injection | 1 | 1 [0 to 0]
  Somnolence Post Injection 1 | 55 | 65 [0 to 0]
  Somnolence Post Injection 2 | 41 | 37 [0 to 0]
  Somnolence Post Injection 3 | 23 | 28 [0 to 0]
  Grade 3 Somnolence Post Any Injection | 2 | 2 [0 to 0]
  Any Anorexia Post Injection 1 | 35 | 42 [0 to 0]
  Anorexia Post Injection 2 | 24 | 22 [0 to 0]
  Anorexia Post Injection 3 | 24 | 25 [0 to 0]
  Grade 3 Anorexia Post Any Injection | 0 | 1 [0 to 0]
  Irritability Post Injection 1 | 85 | 81 [0 to 0]
  Irritability Post Injection 2 | 63 | 65 [0 to 0]
  Irritability Post Injection 3 | 40 | 55 [0 to 0]
  Grade 3 Irritability Post Any Injection | 2 | 1 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 after the first injection to up to 30 days after each injection.
Arm/Group | DTaP-IPV-Hep B-PRP~T Group | Infanrix Hexa™ Group
Serious Adverse Events (participants affected / at risk) | 3/132 | 2/131
Other Adverse Events (participants affected / at risk) | 102/132 | 106/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T Group (N=132) | Infanrix Hexa™ Group (N=131)
Hepatic Cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T Group (N=132) | Infanrix Hexa™ Group (N=131)
Abdominal Pain (Gastrointestinal disorders) | 38 (61) | 44 (65)
Diarrhea (Gastrointestinal disorders) | 17 (19) | 18 (21)
Vomiting (Gastrointestinal disorders) | 29 (29) | 32 (32)
Injection Site Hemorrhage (General disorders) | 8 (9) | 4 (4)
Injection Site Pain (General disorders) | 102 (102) | 101 (101)
Injection Site Erythema (General disorders) | 78 (78) | 66 (66)
Injection Site Swelling (General disorders) | 54 (54) | 52 (52)
Irritability (General disorders) | 100 (100) | 98 (98)
Pyrexia (General disorders) | 37 (37) | 36 (36)
Nasopharyngitis (Infections and infestations) | 62 (78) | 80 (118)
Pharyngitis (Infections and infestations) | 11 (11) | 15 (15)
Anorexia (Infections and infestations) | 54 (54) | 58 (58)
Somnolence (Nervous system disorders) | 73 (73) | 82 (82)
Crying (Psychiatric disorders) | 100 (100) | 93 (93)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 18 (24)
Dermatitis (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 14 (15) | 10 (10)
Pyrexia (General disorders) | 11 (13) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.